CLINICAL TRIAL: NCT00259532
Title: Ultrasound With Contrast Agent, 64-Slice-CT and Tumormarkers for Diagnosing, Evaluation of Operability and Treatment Control of Pancreas Cancer
Brief Title: Three New Methods for Diagnosing Pancreas Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Copenhagen (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: (KF) 01 268342
Record Dates: First submitted 2005-11-25; First posted 2005-11-29 (Estimated); Last update posted 2009-02-26 (Estimated); Status verified 2009-02

CONDITIONS: Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — High-Energy Shock Waves; Contrast Media

INTERVENTIONS:
Procedure: Ultrasound and contrast agent — contrast-enhanced ultrasound combined with the gastrointestinal hormones Secretin and Cholecystokinin, which triggers the enzyme production of pancreas

SUMMARY:
The purpose of this project is to evaluate and compare three new methods for diagnosis, staging, operability evaluation and treatment control of pancreas cancer. The investigators use contrast-enhanced ultrasound combined with the gastrointestinal hormones Secretin and Cholecystokinin, which triggers the enzyme production of pancreas. The hormones induce an increased metabolism and thus an increased blood flow through healthy pancreas tissue, however, not in tumor tissue. The investigators hope to be able to use this effect diagnostically. The patients included will also have a 64-slice-CT in order to evaluate, if an increased diagnostic safety can be reached compared to an older CT scanning method. All patients will also be examined for the tumor marker CA 19-9. Further, the investigators will examine if contrast-enhanced ultrasound can contribute with information in treatment control after either surgery or medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* suspicion of cancer of the pancreas

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2005-02; Study Completion 2009-01

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Nielsen, DMSc, Principal Investigator — Department of Radiology, Section of Ultrasound
Locations (1):
- Copenhagen University Hospital, Copenhagen, Denmark